CLINICAL TRIAL: NCT05808816
Title: Interventional Study on Efficacy of Lactobacillus Crispatus M247 in Patients Affected by HPV Low-grade Preneoplastic Cervical Lesions and Evaluation of Vaginal Microbiota Changes Before and After Oral Supplementation
Brief Title: "Lactobacillus Crispatus M247, LSIL and Microbiota"
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID 4010
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-02

CONDITIONS: Vaginal Flora Imbalance; ASC-US; LSIL; HPV Infection
MeSH Terms: conditions — Atypical Squamous Cells of the Cervix; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Patient with oral supplementation of Lactobacillus Crispatus M247
  Interventions: Drug: Lactobacillus Crispatus M247
- Arm B (No Intervention): Patients without oral supplementation of Lactobacillus Crispatus M247

INTERVENTIONS:
Drug: Lactobacillus Crispatus M247 — Oral supplementation of Lactobacillus Crispatus M247 in patients with cervical low grade lesions HPV related
  Arms: Arm A

SUMMARY:
Patients affected by ASC-US/ low-grade HPV cervical lesions will be randomly assigned to treatment arm vs control arm. The treatment arm will include the characterization of the vaginal microbiota at enrollment (T0), 4 months of oral treatment with Lactobacillus Crispatus M 247 (1 buccal stick Die), characterization of the vaginal microbiota at 1 month post treatment (T5 m). The vaginal microbiota will be evaluated by Danagene microbiome vaginal DNA KIT-XMICROGem (XBIOGem) test, with amplification of the variable regions of the 16S ribosomal RNA gene, using the MICROBIOTA kit (CE-IVD - ARROW diagnostics) and second generation sequencing technologies (NGS on Illumina MiSeq platform). The control arm will provide for the characterization of the vaginal microbiota at the same timescales. Patients will be given a medical history questionnaire at T0 and T5m

ELIGIBILITY:
Inclusion Criteria:

* Pap smear ASCUS or L-SIL
* HPV test + (HPV-HR e/o HPV-LR)

Exclusion Criteria:

* Hormonal therapy (OC, ring, patch, implant)
* Pregnancy status
* Immunosuppressive therapies
* Ongoing HPV vaccination

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of Lactobacillus Crispatus M247 oral supplementation to change the genetic profile of the vaginal microbiota of patients with low-grade lesions from HPV, by XBIOGem test. | 5 months

SECONDARY OUTCOMES:
Cytological regression and microbiological clearance of HPV infection | 5 months
Evaluate the applicability in clinical practice of the XBIOGem test in the characterization of the vaginal microbiota in this type of patient | 24 months
Evaluation of the role of anamnestic factors on the characterization of vaginal microbiota | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, RM, Italy